CLINICAL TRIAL: NCT01183169
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Study on Efficacy and Safety of DEB025 Combined With Peg-IFN Alfa-2a and Ribavirin in Chronic Hepatitis C Genotype 1 Relapsers and Non-responders to Previous Peg-IFN Alfa-2 Plus Ribavirin Treatment
Brief Title: Efficacy and Safety of Adding Alisporivir (DEB025) to Peginterferon (IFN) Alfa-2a (Peg-IFN Alfa-2a) and Ribavirin in Chronic HCV Genotype 1 Patients Who Relapsed or Did Not Respond to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDEB025A2210; 2010-020033-14 (EudraCT Number)
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C
Keywords: Chronic hepatitis C; Cyclophilin inhibitor
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — alisporivir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment A: ALV 600 mg QD (Experimental): Alisporivir (ALV) 600 mg once daily (QD) with Peginterferon alfa-2a (PEG) and Ribavirin (RBV) for up to 48 weeks
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Treatment B: ALV 800 mg QD (Experimental): Alisporivir (ALV) 800 mg QD with PEG and RBV for up to 48 weeks
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Treatment C1: ALV Placebo - 600 mg QD (Experimental): ALV Placebo with PEG and RBV for up to 48 weeks; participants not achieving complete early virologic response (cEVR) after 12 weeks of treatment may switch to active ALV 600 mg QD with PEG and RBV.
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: Placebo
- Treatment C2: ALV Placebo - 400 mg BID (Experimental): ALV Placebo with PEG and RBV for up to 48 weeks; participants not achieving cEVR after 12 weeks of treatment may switch to active ALV 400 mg twice daily (BID) with PEG and RBV.
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: Placebo
- Treatment D: ALV 400 mg BID (Experimental): Alisporivir (ALV) 400 mg twice daily BID with PEG and RBV for up to 48 weeks
  Interventions: Drug: Alisporivir; Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Alisporivir — ALV 200 mg soft gel capsules administered orally
  Other Names: DEB025; ALV
Drug: Peginterferon alfa-2a — PEG 180 μg administered via subcutaneous (s.c.) injection once weekly
  Other Names: Pegasys®; PEG
Drug: Ribavirin — RBV 200 mg tablets (weight-based dose: < 75 mg = 1000 mg/day; ≥ 75 kg = 1200 mg/day) administered orally in a divided daily dose
  Other Names: Copegus®; RBV
Drug: Placebo — ALV placebo soft gel capsules administered orally
  Other Names: ALV Placebo
  Arms: Treatment C1: ALV Placebo - 600 mg QD; Treatment C2: ALV Placebo - 400 mg BID

SUMMARY:
The study is to investigate whether participants with hepatitis C virus (HCV) genotype 1 who have a history of non-response/relapse to peginterferon alfa-2a (PEG) and ribavirin (RBV) may benefit from treatment with triple therapy alisporivir (ALV; DEB025) with PEG and RBV versus placebo with PEG and RBV.

ELIGIBILITY:
Inclusion criteria:

* Chronic HCV genotype 1 viral infection
* HCV RNA ≥ 1,000 IU/ml assessed by quantitative polymerase chain reaction (qPCR) or equivalent at screening
* Previous non-responders/relapsers to PEG and RBV after treatment for at least 12 weeks

Exclusion criteria:

* Treatment with any anti-HCV drug (whether approved or investigational) within 3 months prior to screening
* Women of child-bearing potential unless using highly effective
* Any other cause of relevant liver disease other than HCV
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (67):
- United States (16):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Egg Harbor Twp, New Jersey
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Australia (5):
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- France (2):
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
- Hungary (5):
  - Novartis Investigative Site, Békéscsaba
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Székesfehérvár
- Italy (6):
  - Novartis Investigative Site, Antella - Bagno A Ripoli, FI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Bologna
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Lódz
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Romania (5):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Iași, Iaşi
  - Novartis Investigative Site, Bucharest, Romania
  - Novartis Investigative Site, Bucharest
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
- Taiwan (7):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Douliu
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Keelung
  - Novartis Investigative Site, Lin-Ko
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Fatih / Istanbul
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: Alisporivir (ALV; DEB025) 600 mg once daily (QD) with peginterferon alfa-2a (PEG) and ribavirin (RBV) for up to 48 weeks.
- Treatment B: ALV 800 mg QD with PEG and RBV for up to 48 weeks.
- Treatment C1: Treatment C subset C1: ALV placebo with PEG and RBV for up to 48 weeks; participants not achieving complete early virologic response (cEVR: hepatitis C virus (HCV) ribonucleic acid (RNA) <LOQ after 12 weeks of treatment) could switch to active ALV 600 mg QD with PEG and RBV.
- Treatment C2: Treatment C subset C2: ALV placebo with PEG and RBV for up to 48 weeks; participants not achieving cEVR could switch to active ALV 400 mg twice daily (BID) with PEG and RBV.
- Treatment D: ALV 400 mg BID with PEG and RBV for up to 48 weeks.
- Treatment C1A: ALV 600 mg QD with PEG and RBV in participants not achieving cEVR in Treatment C subset C1.
- Treatment C2A: ALV 400 mg BID with PEG and RBV in participants not achieving cEVR in Treatment C subset C2.
Period: Main Phase
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment C1A | Treatment C2A
Started | 121 | 115 | 59 | 55 | 109 | 0 | 0
Completed Treatment | 72 | 78 | 17 | 17 | 77 | 0 | 0
Switched to ALV | 0 | 0 | 35 | 30 | 0 | 0 | 0
Completed | 94 | 93 | 18 | 18 | 83 | 0 | 0
Not Completed | 27 | 22 | 41 | 37 | 26 | 0 | 0
Period: Post-switch Phase
Arm/Group | Treatment A | Treatment B | Treatment C1 | Treatment C2 | Treatment D | Treatment C1A | Treatment C2A
Started | 0 (Not a post-switch group) | 0 (Not a post-switch group) | 0 (Not a post-switch group) | 0 (Not a post-switch group) | 0 (Not a post-switch group) | 35 (Participants in Treatment C1 who switched to active ALV) | 30 (Participants in Treatment C2 who switched to active ALV)
Completed Treatment | 0 | 0 | 0 | 0 | 0 | 12 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 21 | 21
Not Completed | 0 | 0 | 0 | 0 | 0 | 14 | 9

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Treatment A: ALV 600 mg QD with PEG and RBV for up to 48 weeks.
- Treatment C: Treatment C1 + Treatment C2. ALV placebo with PEG and RBV for up to 48 weeks; participants not achieving cEVR could switch to active ALV.
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Total
Number analyzed (Participants) | 121 | 115 | 114 | 109 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.24) | 50.9 (10.11) | 50.5 (10.50) | 51.0 (9.68) | 50.6 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 47 | 36 | 40 | 181
  Male | 63 | 68 | 78 | 69 | 278

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Early Viral Response Below the Limit of Quantification (cEVR-LOQ)
Description: cEVR-LOQ was defined as serum HCV RNA below the limit of quantification (< LOQ; i.e., 25 IU/mL) after 12 weeks of treatment. Post-switch groups were assessed 12 weeks after the switch.
Time Frame: after 12 weeks of treatment
Population: Full Analysis Set (FAS) For Efficacy, defined as all randomized participants who were randomized after the 2nd protocol amendment
Measure: Number; unit: percentage of participants
Groups:
- Treatment C: ALV placebo with PEG and RBV for up to 48 weeks; participants not achieving cEVR could switch to active ALV.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants | 48.2 | 61.1 | 35.5 | 74.3 | 45.5 | 80.0

2. Secondary Outcome: Percentage of Participants With Complete Early Viral Response Below the Limit of Detection (cEVR-LOD)
Description: cEVR-LOD was defined as serum HCV RNA below the limit of detection (< LOD; i.e., 10 IU/mL) after 12 weeks of treatment. Post-switch groups were assessed 12 weeks after the switch.
Time Frame: after 12 weeks of treatment
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants | 39.1 | 41.7 | 20.9 | 58.7 | 39.4 | 73.3

3. Secondary Outcome: Percentage of Participants Who Achieved Sustained Viral Response 12 Weeks After Treatment (SVR12)-LOQ and SVR12-LOD
Description: SVR12-LOQ and SVR12-LOD were defined as serum HCV RNA < LOQ and serum HCV RNA < LOD 12 weeks after treatment, respectively.
Time Frame: 12 weeks after treatment
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants
  SVR12-LOQ | 42.7 | 51.9 | 14.5 | 65.1 | 18.2 | 53.3
  SVR12-LOD | 40.9 | 50.9 | 14.5 | 63.3 | 18.2 | 53.3

4. Secondary Outcome: Percentage of Participants Who Achieved Sustained Viral Response 24 Weeks After Treatment (SVR24)-LOQ and SVR24-LOD
Description: SVR24-LOQ and SVR24-LOD were defined as serum HCV RNA < LOQ and serum HCV RNA < LOD 24 weeks after treatment, respectively.
Time Frame: 24 weeks after treatment
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants
  SVR24-LOQ | 41.8 | 51.9 | 14.5 | 65.1 | 18.2 | 53.3
  SVR24-LOD | 40.0 | 50.0 | 14.5 | 63.3 | 18.2 | 53.3

5. Secondary Outcome: Percentage of Participants With Rapid Viral Response (RVR)-LOQ and RVR-LOD
Description: RVR-LOQ and RVR-LOD were defined as serum HCV RNA < LOQ and serum HCV RNA < LOD after 4 weeks of treatment, respectively. Post-switch groups were assessed 4 weeks after the switch.
Time Frame: after 4 weeks of treatment
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants
  RVR-LOQ | 20.9 | 25.0 | 7.3 | 41.3 | 39.4 | 56.7
  RVR-LOD | 9.1 | 8.3 | 2.7 | 22.9 | 18.2 | 50.0

6. Secondary Outcome: Percentage of Participants With Partial Early Virologic Response After 12 Weeks of Treatment (pEVR)-LOQ and pEVR-LOD
Description: pEVR-LOQ and pEVR-LOD were defined as a ≥ 2 log10 decrease in HCV RNA and still detectable (≥ LOQ and ≥ LOD, respectively) after 12 weeks of treatment. Post-switch groups were assessed 12 weeks after the switch.
Time Frame: after 12 weeks of treatment
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants
  pEVR-LOQ | 38.2 | 28.7 | 31.8 | 11.9 | 3.0 | 6.7
  pEVR-LOD | 47.3 | 48.1 | 46.4 | 27.5 | 9.1 | 13.3

7. Secondary Outcome: Percentage of Participants With End of Treatment Response (ETR)-LOQ and ETR-LOD
Description: ETR-LOQ and ETR-LOD were defined as serum HCV RNA < LOQ and serum HCV RNA < LOD at treatment end (completed or prematurely discontinued), respectively.
Time Frame: within 48 weeks
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants
  ETR-LOQ | 68.2 | 74.1 | 33.6 | 82.6 | 51.5 | 73.3
  ETR-LOD | 61.8 | 70.4 | 31.8 | 78.9 | 36.4 | 66.7

8. Secondary Outcome: Percentage of Participants With Abnormal Alanine Aminotransferase (ALT) at Baseline Who Had Normalized ALT at Treatment End and Study End
Time Frame: Up to 48 weeks
Population: Participants in the FAS For Efficacy with abnormal ALT at baseline and available data at the respective time point
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 53 | 49 | 61 | 53 | 14 | 7
percentage of participants
  End of Treatment (n = 53,49,60,53,14,7) | 77.4 | 77.6 | 59.0 | 83.0 | 35.7 | 28.6
  End of Study (n = 49,42,18,46,13,6) | 54.7 | 61.2 | 18.0 | 67.9 | 21.4 | 28.6

9. Secondary Outcome: Percentage of Participants With On-treatment Viral Breakthrough
Description: On-treatment viral breakthrough was defined as either:
  * Confirmed increase of HCV RNA ≥1 log10 above nadir (nadir = lowest HCV RNA value during treatment), or
  * HCV RNA becoming ≥ 100 IU/mL after previously being undetectable (< LOQ) during treatment
Time Frame: within 48 weeks
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants | 12.7 | 9.3 | 5.5 | 2.8 | 6.1 | 10.0

10. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as reappearance of detectable HCV RNA after previously being undetectable (< LOQ) during treatment.
Time Frame: within 24 weeks after treatment
Population: FAS For Efficacy
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment C1A | Treatment C2A
Number analyzed (Participants) | 110 | 108 | 110 | 109 | 33 | 30
percentage of participants | 19.1 | 18.5 | 17.3 | 12.8 | 30.3 | 13.3

ADVERSE EVENTS:
Groups:
- Treatment A: On-treatment AEs: Adverse events (AEs) occurring while on treatment in participants receiving ALV 600 mg QD with PEG and RBV for up to 48 weeks.
- Treatment B: On-treatment AEs: AEs occurring while on treatment in participants receiving ALV 800 mg QD with PEG and RBV for up to 48 weeks.
- Treatment C1: On-treatment AEs; Treatment C1: Post-treatment AEs: AEs occurring while on treatment in participants receiving ALV placebo (and may have received ALV 600 mg QD post-switch) with PEG and RBV for up to 48 weeks.
- Treatment C2: On-treatment AEs; Treatment C2: Post-treatment AEs: AEs occurring while on treatment in participants receiving ALV placebo (and may have received ALV 400 mg BID post-switch) with PEG and RBV for up to 48 weeks.
- Treatment D: On-treatment AEs: AEs occurring while on treatment in participants receiving ALV 400 mg BID with PEG and RBV for up to 48 weeks.
- Treatment A: Post-treatment AEs: AEs occurring after end of treatment in participants receiving ALV 600 mg QD with PEG and RBV for up to 48 weeks.
- Treatment B: Post-treatment AEs: AEs occurring after end of treatment in participants receiving ALV 800 mg QD with PEG and RBV for up to 48 weeks.
- Treatment D: Post-treatment AEs: AEs occurring after end of treatment in participants receiving ALV 400 mg BID with PEG and RBV for up to 48 weeks.
Arm/Group | Treatment A: On-treatment AEs | Treatment B: On-treatment AEs | Treatment C1: On-treatment AEs | Treatment C2: On-treatment AEs | Treatment D: On-treatment AEs | Treatment A: Post-treatment AEs | Treatment B: Post-treatment AEs | Treatment C1: Post-treatment AEs | Treatment C2: Post-treatment AEs | Treatment D: Post-treatment AEs
Serious Adverse Events (participants affected / at risk) | 7/120 | 11/115 | 5/59 | 1/55 | 18/108 | 2/120 | 4/115 | 0/59 | 0/55 | 0/108
Other Adverse Events (participants affected / at risk) | 116/120 | 108/115 | 58/59 | 54/55 | 106/108 | 22/120 | 21/115 | 13/59 | 10/55 | 19/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: On-treatment AEs (N=120) | Treatment B: On-treatment AEs (N=115) | Treatment C1: On-treatment AEs (N=59) | Treatment C2: On-treatment AEs (N=55) | Treatment D: On-treatment AEs (N=108) | Treatment A: Post-treatment AEs (N=120) | Treatment B: Post-treatment AEs (N=115) | Treatment C1: Post-treatment AEs (N=59) | Treatment C2: Post-treatment AEs (N=55) | Treatment D: Post-treatment AEs (N=108)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug interaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: On-treatment AEs (N=120) | Treatment B: On-treatment AEs (N=115) | Treatment C1: On-treatment AEs (N=59) | Treatment C2: On-treatment AEs (N=55) | Treatment D: On-treatment AEs (N=108) | Treatment A: Post-treatment AEs (N=120) | Treatment B: Post-treatment AEs (N=115) | Treatment C1: Post-treatment AEs (N=59) | Treatment C2: Post-treatment AEs (N=55) | Treatment D: Post-treatment AEs (N=108)
Anaemia (Blood and lymphatic system disorders) | 49 | 41 | 24 | 21 | 51 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 17 | 13 | 8 | 6 | 20 | 0 | 0 | 3 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 2 | 4 | 0 | 8 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 49 | 40 | 22 | 16 | 46 | 0 | 0 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 19 | 4 | 6 | 28 | 1 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 11 | 7 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 2 | 3 | 5 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 4 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 7 | 6 | 2 | 7 | 14 | 2 | 0 | 1 | 1 | 1
Dry eye (Eye disorders) | 7 | 7 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 5 | 8 | 1 | 3 | 14 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 4 | 8 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 5 | 2 | 2 | 7 | 1 | 0 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 7 | 7 | 6 | 6 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 15 | 8 | 5 | 5 | 13 | 0 | 1 | 2 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 6 | 3 | 3 | 2 | 6 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 6 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 10 | 7 | 2 | 5 | 15 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 19 | 18 | 11 | 9 | 10 | 0 | 0 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 15 | 10 | 5 | 8 | 10 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 15 | 4 | 5 | 2 | 15 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 7 | 10 | 3 | 5 | 3 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 46 | 35 | 17 | 17 | 51 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 19 | 18 | 7 | 9 | 19 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 19 | 30 | 9 | 14 | 17 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 3 | 4 | 2 | 6 | 4 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 14 | 13 | 6 | 5 | 14 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 47 | 45 | 25 | 27 | 45 | 1 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 13 | 10 | 15 | 6 | 11 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 8 | 11 | 5 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 8 | 7 | 3 | 3 | 6 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 9 | 8 | 2 | 2 | 9 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 32 | 34 | 18 | 18 | 28 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 19 | 14 | 4 | 6 | 36 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 14 | 11 | 5 | 6 | 18 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 5 | 1 | 3 | 4 | 0 | 1 | 0 | 0 | 3
Oral herpes (Infections and infestations) | 4 | 7 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 3 | 2 | 2 | 6 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 5 | 3 | 6 | 6 | 1 | 0 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 7 | 2 | 4 | 3 | 9 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 1 | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 2
Lipase increased (Investigations) | 2 | 1 | 4 | 2 | 5 | 0 | 0 | 0 | 0 | 0
Total bile acids increased (Investigations) | 5 | 3 | 3 | 1 | 8 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 9 | 9 | 3 | 4 | 9 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 31 | 23 | 9 | 12 | 26 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 | 21 | 4 | 3 | 18 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 19 | 8 | 8 | 9 | 2 | 1 | 1 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 5 | 4 | 6 | 10 | 2 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 12 | 3 | 5 | 17 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 21 | 16 | 13 | 18 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 0 | 2 | 6 | 2 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5 | 3 | 1 | 5 | 1 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 9 | 10 | 3 | 5 | 4 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 20 | 22 | 11 | 8 | 15 | 0 | 1 | 1 | 2 | 4
Dysgeusia (Nervous system disorders) | 5 | 7 | 4 | 5 | 9 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 59 | 47 | 24 | 22 | 38 | 2 | 2 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 6 | 2 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 5 | 4 | 2 | 6 | 3 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 19 | 8 | 4 | 5 | 11 | 2 | 1 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 3 | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 22 | 14 | 10 | 7 | 13 | 0 | 2 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 35 | 24 | 11 | 19 | 17 | 1 | 2 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 1 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 7 | 4 | 2 | 4 | 1 | 1 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 4 | 4 | 1 | 2 | 0 | 0 | 2 | 0 | 0
Suspiciousness (Psychiatric disorders) | 1 | 4 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 29 | 18 | 17 | 16 | 2 | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 8 | 6 | 5 | 16 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 3 | 6 | 8 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4 | 2 | 10 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 5 | 4 | 8 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 23 | 10 | 9 | 19 | 0 | 1 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 16 | 11 | 12 | 16 | 1 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 6 | 7 | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 5 | 2 | 3 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 30 | 21 | 17 | 32 | 2 | 2 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 23 | 22 | 15 | 9 | 17 | 3 | 2 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 21 | 22 | 5 | 11 | 28 | 2 | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
In April 2012, ALV and placebo were discontinued in all participants. Participants remained on PEG and RBV treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other